CLINICAL TRIAL: NCT02962622
Title: Soluble Insulin Receptor Dysfunction Correlates With HAND in HIV+ Women on CART
Brief Title: Cognition Metabolism and Exercise Among Women Living With HIV in Puerto Rico
Acronym: CMEx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Puerto Rico (Other)
Responsible Party: Principal Investigator, Farah A. Ramirez-Marrero, Professor, University of Puerto Rico
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: UPuertoRico
Record Dates: First submitted 2016-10-05; First posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: HIV
Keywords: Neurocognition; Exercise; Metabolism; Hispanic women
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hispanic women living with HIV (Experimental): High intensity interval training (HIIT) on normally active but physically untrained HIV+ Hispanic women, one with (n=15) and other without (n=15) neuro-cognitive impairment (HAND) on antiretroviral therapy (CART) receive 2 weeks, 6 sessions of 8 x 60 seconds cycling bouts eliciting approximately 80% of maximal heart rate with 60 second rest between bouts after which they will receive 4 week, 12 sessions of 10 x 60 seconds cycling bouts eliciting approximately 90% of maximal heart rate with 60 second rest between bouts.
  Interventions: Other: High intensity interval training (HIIT)
- Hispanic women living without HIV (Experimental): High intensity interval training (HIIT) on a comparison group of 15 Hispanic women without HIV receive 2 weeks, 6 sessions of 8 x 60 seconds cycling bouts eliciting approximately 80% of maximal heart rate with 60 second rest between bouts after which they will receive 4 week, 12 sessions of 10 x 60 seconds cycling bouts eliciting approximately 90% of maximal heart rate with 60 second rest between bouts.
  Interventions: Other: High intensity interval training (HIIT)

INTERVENTIONS:
Other: High intensity interval training (HIIT) — Six weeks, three days per week (total of 18 sessions) of HIIT cycle ergometer exercise protocol

SUMMARY:
The study evaluates the association between soluble insulin receptor dysfunction, cardiorespiratory fitness, and HIV associated neurocognitive disorder (HAND). Those who volunteer to participate in the study will have two evaluations at study entry that include a dual x-ray absorptiometry (DEXA) densitometry, anthropometry, neurocognitive testing, blood and urine samples for metabolic testing, and a cardiorespiratory fitness testing. DEXA will be conducted in the Endocrinology Unit at the University Hospital, Medical Center (letter of support included). The cardiorespiratory fitness testing will be conducted in the AIDS Clinical Trials Unit (ACTU) project, University of Puerto Rico, Medical Sciences Campus, and the Puerto Rico Clinical and Translational Research Consortium. Then, participants will be invited to participate in a 6-week, 3 days/week individualized exercise program. The exercise program will be conducted at the University of Puerto Rico Medical Sciences Campus. After completion of the exercise program, study entry evaluations will be repeated. The duration of the study will take approximately 10 weeks.

DETAILED DESCRIPTION:
The aim of the study is to determine the effect of a low volume high intensity interval training (HIIT) exercise intervention on cardio-respiratory fitness (CR-fitness), insulin resistance, and cognitive function among normally active but physically untrained HIV+ Hispanic women. The primary hypotheses are that HIIT will improve: 1) CR-fitness in all groups (HIV+ and HIV-), 2) insulin sensitivity in both groups of HIV+ women, and 3) cognitive function as determined by hippocampal function in HIV+ women with HAND. Participants will receive 2 weeks, 6 sessions of 8 x 60 seconds cycling bouts eliciting approximately 80% of maximal heart rate with 60 second rest between bouts after which they will receive 4 week, 12 sessions of 10 x 60 seconds cycling bouts eliciting approximately 90% of maximal heart rate with 60 second rest between bouts. Then, participants will be evaluated with a CR-fitness, insulin resistance, anthropometry, and neurocognitive function tests.

Participants will undergo an intervention (described above) designed for normally active but physically untrained HIV+ Hispanic women, one with (n=15) and other without (n=15) neurocognitive impairment & HIV- controls (n=15). After the HIIT intervention, measurements of CR-fitness, insulin resistance, and cognitive function including hippocampal function using the memory island test will be obtained, as well as CR-fitness, anthropometry, DEXA densitometry, and blood and urine samples for metabolic testing. The ultimate goal is to improve the understanding of mechanisms by which exercise influence neurocognitive function; thus, providing a potential non-pharmacological alternative to prevent, control or reduce chronic incapacitating diseases in HIV+ Hispanic adults.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-seropositive women ≥21 years with lymphocytes differentiated cells 4 (CD4) cell count or nadir in the last year ≤500 cells/mm3, or viral load ≥1,000 copies/mL despite highly active antiretroviral therapy (HAART).
2. Education level ≥9th grade, since is the minimum required for some of the neuro-psychological (NP) tests. All HIV-seropositive and HIV-seronegative participants will be tested for vocabulary and reading pre-morbid cognitive function as described below.
3. Non-drug abusers; defined as those with <5 exposures in a lifetime to drugs (opiates/heroin, methamphetamine, cocaine/crack, speed ball). For the purpose of this study neither tobacco nor nicotine use will be considered a drug.
4. No diagnosis of diabetes or the use of hypoglycemic agents.

Exclusion Criteria:

1. HIV+ women and men <21 years old with CD4 cell count >500 cells/mm3 and/or viral load <1,000 copies/mL.
2. Opportunistic infections of the central nervous system (CNS) as determined by neurological evaluation and neuroimaging. (Neuroimaging studies, if needed, will be performed as part of patient care and hence have not been included as a budget item in this proposal.)
3. History of diabetes or the use hypoglycemic agents.
4. Underlying neurologic and/or neuropsychiatric disorders such as cerebrovascular events; history of meningitis/encephalitis, CNS opportunistic infections, or seizures; head trauma (<6 months with loss of consciousness for >1 hr); cerebral palsy; or any other neuropsychiatric condition that in the judgment of the investigators may affect the study.
5. Active systemic infection or illness, which in the judgment of the investigators may affect the study.
6. Pregnant/nursing mothers or women with recent birth (<60 days).
7. Substance abuse: active drug use - all participants will be screened with urine toxicology and active alcohol abuse - those scoring >3 points in the Michigan Alcoholism Screening Test (MAST) will be screened with blood samples for alcohol levels (Seltzer 1975).
8. Patients who are unwilling to give informed consent or incapable of understanding informed consent.
9. Education less than 9th grade.

   -

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Cardio-respiratory fitness as measured by maximal oxygen consumption (VO2max) | 6 weeks
  Maximal oxygen consumption

SECONDARY OUTCOMES:
Metabolic syndrome classification based on the National Cholesterol Education Program (NCEP) criteria | 6 weeks
  Number of participants with abnormal values in 3 or more of the following: fasting glucose, resting blood pressure, waist circumference, fasting triglycerides, and HDL.
Neurocognitive function as measured by memory testing | 6 weeks
  Number of participants with abnormal values of neurocognitive function will be identified. Measures of memory testing using questionnaires and a computer-based assessment will be aggregated to arrive at one reported value of neurocognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Farah A. Ramirez-Marrero, PhD, Principal Investigator — University of Puerto Rico
Locations (1):
- Medical Sciences Campus, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ramirez-Marrero FA, Perez-Frontera S, Amalbert-Birriel MA, Matos M, Santana-Bagur J, Frontera WR, Wojna V. Brief Report: Effects of Low-Volume High-Intensity Interval Training in Hispanic HIV+ Women: A Nonrandomized Study. J Acquir Immune Defic Syndr. 2020 Jul 1;84(3):285-289. doi: 10.1097/QAI.0000000000002353. PMID 32530906